CLINICAL TRIAL: NCT00132652
Title: A Randomized Trial of Switching Antiviral Therapy From Lamivudine to Telbivudine (LdT) vs. Continued Lamivudine Treatment in Adults With Chronic Hepatitis B
Brief Title: Switching Therapy From Lamivudine to Telbivudine Versus Continued Lamivudine in Adults With Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV-02B-019
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; Telbivudine

INTERVENTIONS:
Drug: Lamivudine
Drug: Telbivudine

SUMMARY:
This study is being conducted to compare the safety and effectiveness of switching treatment from lamivudine to telbivudine (LdT) against continued lamivudine treatment. Results from patients who were taking lamivudine and then switched to telbivudine will be compared with the results from patients who continued on lamivudine alone.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical history compatible with chronic hepatitis B
* Patient has compensated liver disease
* Patient has received previous treatment with lamivudine for a duration of at least 3 months and not more than 12 months

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient is co-infected with hepatitis C, hepatitis D or HIV
* Patient previously received antiviral treatment for hepatitis B other than lamivudine in the preceding 12 months

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (3):
  - San Diego, California
  - New York, New York
  - Philadelphia, Pennsylvania
- Westmead, Australia
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Beijing, China
- Nice, France
- Tel Aviv, Israel
- Auckland, New Zealand
- Singapore, Singapore
- Tainan, Taiwan
- Chiang Mai, Thailand
- London, United Kingdom

REFERENCES:
- See also: Related Info — http://onlinelibrary.wiley.com/doi/10.1111/j.1478-3231.2010.02360.x/pdf